CLINICAL TRIAL: NCT02642016
Title: A Phase 1, Open-label, Dose-escalation and Expansion Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of CDX-0158 in Adult Patients With KIT Positive Advanced Solid Tumors.
Brief Title: A Study to Evaluate the Safety and Pharmacokinetics of CDX-0158 in Adult Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDX0158-CL-001
Record Dates: First submitted 2015-12-16; First posted 2015-12-30 (Estimated); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Advanced Cancer
Keywords: KTN0158; Advanced Cancer; Phase 1; Monoclonal Antibody; Safety and Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CDX-0158 (Experimental)
  Interventions: Biological: CDX-0158 (formerly known as KTN-0158)

INTERVENTIONS:
Biological: CDX-0158 (formerly known as KTN-0158) — Single agent CDX-0158 until unacceptable toxicity or progressive disease

SUMMARY:
This is a dose-escalation Phase 1 study designed to determine the maximum tolerated dose (MTD) and/or recommended Phase 2 dose, and the safety profile of CDX-0158 in patients with KIT-positive advanced solid malignancies refractory to standard therapy or for which no standard therapy exists.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and any locally required authorization (eg, HIPAA) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
2. Metastatic or unresectable cancer that expresses KIT as documented in the patient's pathology report.
3. For patients with GIST, patients will have progressed on at least one prior tyrosine kinase inhibitor therapy or be intolerant. If documented to have SDH deficient or PDGFRA-D842V GIST, no prior therapy is required for study entry. Other patients with KIT positive cancers will have progressed on at least one prior therapy.
4. Patients must have at least 1 lesion that is measurable using RECIST guidelines.
5. Females of childbearing potential who are sexually active with a nonsterilized male partner must use 2 methods of effective contraception from screening, and must agree to continue using such precautions for 60 days after the final dose of study medication. Females of childbearing potential are defined as those who are not surgically sterile (i.e., bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or those who are postmenopausal (defined as 12 months with no menses without an alternative medical cause).
6. Nonsterilized males who are sexually active with a female partner of childbearing potential must, with their partner, use 2 acceptable methods of effective contraception from Day 1 through 60 days after receipt of the final dose of study medication.
7. ECOG status of 0 or 1.
8. Adequate organ function as defined below:

   * Hemoglobin ≥ 9 g/dL. This criterion must be met without transfusion.
   * Absolute neutrophil count ≥ 1500/mm3
   * Platelet count ≥ 100,000/mm3
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5 × upper limit of normal (ULN) for cases involving liver metastasis and ≤ 2.5 ×ULN for all other cases
   * Bilirubin ≤ 1.5 × ULN except for cases of documented or suspected Gilbert's disease, in which bilirubin must be ≤ 5 × ULN
   * Serum creatinine ≤ 1.5 g/dL

Exclusion Criteria:

1. Receipt of anticancer therapy:

   * Within 3 weeks prior to the first dose of CDX-0158 of any biologic treatment or IV chemotherapy.
   * Within 2 weeks prior to the first dose of CDX-0158 of any oral therapy or 5.5 half lives whichever is longer or following palliative radiation therapy.

   Concurrent use of hormones for non-cancer related conditions (e.g., insulin for diabetes and hormone replacement therapy) is acceptable.
2. Requirement for chronic immunosuppressive medication including systemic corticosteroids above the physiologic dose (30 mg/day hydrocortisone or the equivalent).
3. Known allergy or past administration reaction including infusion related reaction (IRRs), anaphylactic, or anaphylactoid reactions to any component of the CDX-0158 formulation.
4. History of clinically significant allergic reactions or atopic disease that may pose an increased risk of severe CDX-0158 IRRs.
5. Symptomatic or untreated central nervous system metastases requiring concurrent treatment, including but not limited to surgery, radiation, and/or corticosteroids; if treated, patient must be asymptomatic for 3 months prior to study entry.
6. Other invasive malignancy within 2 years prior to enrollment (localized prostate cancer, cervical carcinoma in situ, non-melanoma skin cancer, or ductal carcinoma in situ of the breast that has/have been surgically cured would not be exclusionary).
7. Unresolved toxicities from prior anticancer therapy, defined as having not resolved to NCI CTCAE v 4.03 < Grade 2 or normalized to baseline, or to levels dictated in the inclusion/exclusion criteria, with the exception of alopecia.
8. Major surgical procedure (as defined by the investigator) within 30 days prior to Study Day 1 or incomplete recovery from any prior surgery.
9. Pregnancy or breast feeding
10. Uncontrolled intercurrent illness that would limit compliance with study requirements or compromise the patient such as ongoing or active infection, symptomatic congestive heart failure, hypertension requiring adjustment of medication, idiopathic and symptomatic hypotension, unstable angina pectoris, clinically significant cardiac arrhythmia including uncontrolled atrial fibrillation, active peptic ulcer disease or gastritis with ongoing blood loss, or psychiatric illness/social situations that would limit compliance or compromise the ability of the patient to give written informed consent.
11. Any condition that, in the opinion of the investigator, would interfere with evaluation of the study medication or interpretation of patient safety or study results.
12. Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) study.
13. Patients with a left ventricular cardiac ejection fraction < 50% as assessed by an echocardiogram or MUGA scan or prolonged QTc interval of Grade 2 or higher or history of prolonged QTc interval from other drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-12; Primary Completion 2018-01-30 (Actual); Study Completion 2019-06-04 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities for CDX-0158 | Participants will be evaluated for DLTs from the first adminstration of CDX-0158 through 21 days following initial dosing.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Oregon Health & Sciences University, Portland, Oregon
  - Sarah Cannon Research Institute, Nashville, Tennessee